CLINICAL TRIAL: NCT06148155
Title: A Study of [68Ga]Ga-NOTA-RG2 PET Imaging in the Diagnosis of Hepatocellular
Brief Title: A Study of [68Ga]Ga-NOTA-RG2 PET Imaging in the Diagnosis of Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-544
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Positron-Emission Tomography
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with primary and/or metastatic hepatocellular carcinoma (HCC) (Experimental): The diagnosis of HCC is established by surgery or biopsy pathology.
  Interventions: Radiation: [68Ga]Ga-NOTA-RG2 PET Imaging

INTERVENTIONS:
Radiation: [68Ga]Ga-NOTA-RG2 PET Imaging — Intravenous injection of 1.8 MBq [0.05MCi]/kg of [68Ga]Ga-NOTA-RG2 in a single dose.

SUMMARY:
The aim of this study was to establish and optimize the imaging method of [68Ga]Ga-NOTA-RG2, as well as its physiological and pathological distribution characteristics, and on this basis to evaluate the diagnostic efficacy of the above imaging agents in patients with hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma patients

  1. Age between 18 and 65 years old, gender is not limited.
  2. Patients with suspicious intrahepatic spaces detected by MR and considered to be hepatocellular carcinoma with AFP>200 ug/L who have not undergone surgery.
  3. Patients with hepatocellular carcinoma confirmed by puncture pathology
  4. Written informed consent must be signed by the subject or his/her legal guardian or caregiver.
  5. Willingness and ability to cooperate with all programs of the study.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Patients receiving anti-tumor therapy prior to the PET/CT scan.
  2. Suffering from severe other neurological disorders, or gastrointestinal, cardiovascular, hepatic, renal, hematologic, respiratory, immunodeficiency, and other serious diseases.
  3. Alternative subjects with conditions that contraindicate PET/CT scanning. This includes, but is not limited to, elevated blood glucose that is not effectively controlled; pregnant, lactating, or breastfeeding women; those who are unable to receive repeated intravenous injections; those who may be hypersensitive to the drug and its components (including a history of severe allergies or anaphylactic reactions, especially to the drug being examined); and hermetic phobias.
  4. Within the past year, have participated in other research protocols or clinical care, in addition to the radiation exposure expected from participation in this clinical study, which has resulted in radiation exposure in excess of an effective dose of 50 mSv.
  5. Alternative subjects have undergone major surgery within the last 3 months; experimental drug or device therapy (of uncertain efficacy or safety) within 1 month
  6. The alternate subject has any clinical condition that, in the opinion of the Sponsor of this study, may cause or has the potential to cause harm from this agent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Complete PET imaging | 90mins from time of injection
  To assess the sensitivity and specificity of diagnosing HCC using [68Ga]Ga-NOTA-RG2.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China